CLINICAL TRIAL: NCT07139080
Title: The Effect of Mobile Application-Based Education on Self-Efficacy, Medication Adherence and Sleep Quality in Asthma Patients.
Brief Title: Effect of Mobile Application-Based Education on Self-Efficacy, Medication Adherence and Sleep Quality in Asthma.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gulhane Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Ezgi Yildirim, Principal İnvestigator, Gulhane Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Asthma Mobil Nursing Education
Record Dates: First submitted 2025-05-08; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: PATIENT EDUCATION
Keywords: Asthma; Self Efficacy; Medication Adherence; Mobile Education; Sleep
MeSH Terms: conditions — Asthma; Medication Adherence

STUDY DESIGN:
Who Masked: Participant
Masking Description: Randomization will be performed according to disease duration via calculatorsoup.com, a web-based program. It will be defined as the intervention group (M) and the control group (K). During the randomization process, numbered envelopes will be prepared by an academician outside the research for the patients included in the intervention and control groups. The researcher will learn the information about the intervention or control group in the prepared envelopes when the relevant envelope is opened during the interview with the patient. Thus, statistical blinding will be ensured.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile Education Group (Experimental): It consists of participants who will download the mobile patient education and breathing exercise reminder program and apply it for 10 weeks.
  Interventions: Behavioral: Mobile education
- Control Group (No Intervention): This is the group of participants to be followed within the standard treatment plan. A mobile training and breathing exercise reminder program will be downloaded to patients in this group at the end of the study.

INTERVENTIONS:
Behavioral: Mobile education — It consists of participants who will download the mobile patient education and breathing exercise reminder program and apply it for 10 weeks.
  Arms: Mobile Education Group

SUMMARY:
Asthma patients with recurrent airway obstruction frequently exhibit poor symptom control, characterized by treatment non-adherence and sleep-wake cycle disturbances. A nurse-led mobile health education intervention may address these challenges by enhancing collaborative disease management, enabling remote patient monitoring, and strengthening self-management competencies.

The AstımAsistan application was designed to monitor changes in patient self-efficacy, medication adherence, and sleep quality through three core features: (1) patient education modules, (2) breathing exercise/medication reminders, and (3) mobile consultation capabilities.

Study data were collected using four instruments: (1) the Participant Information Form, (2) the Chronic Disease Self-Efficacy Scale, (3) the Medication Adherence Reporting Scale, and (4) the Pittsburgh Sleep Quality Index. The mobile education-based application was developed following the ADDIE (Analysis, Design, Development, Implementation, and Evaluation) instructional design model."

ELIGIBILITY:
Inclusion Criteria:

1. Being between the ages of 18-65
2. Having been diagnosed with asthma at least 6 months ago
3. Being treated for asthma in oral, inhaler or injection forms
4. Being literate in Turkish
5. Having an Android phone on which the mobile application can be installed and being able to use the phone
6. Having mobile network or wireless internet access
7. Volunteering to participate in research
8. Living in Ankara

Exclusion Criteria:

1. Being hospitalized for asthma treatment
2. Having a language barrier that hinders communication
3. Being diagnosed with COPD
4. Being diagnosed with a psychiatric disease
5. Being on psychoactive or opioid therapy
6. Being diagnosed with a sleep disorder related to non-respiratory reasons (physical and psychological) and being treated

Exclusion criteria when the study is going on :

Intervention group;

1. The participant was diagnosed with a health problem requiring inpatient treatment during the study period.
2. The participant withdraws from the study voluntarily.
3. Inability to use the mobile application during the research
4. Reading fewer than 6 theme headings in the mobile application (75% or less) and missing breathing exercises for more than 16 days (80% or less)

Control group;

1. The participant was diagnosed with a health problem requiring inpatient treatment during the study period.
2. The participant withdraws from the study voluntarily.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-04-28 (Actual); Study Completion 2025-04-28 (Actual)

PRIMARY OUTCOMES:
Chronic Disease Self-Efficacy | 10 weeks
  Chronic Disease Self Efficacy Scale: In this 30-item scale, each question is scored between 1 and 10 points to determine the level of self-efficacy. The total score obtained by the individual from the scale is divided by the number of items to calculate an overall self-efficacy average. The scale also has 10 subtitles. If the 30 items' average is below 7, it means the individual has low self-efficacy. If the average is 7 or above, it indicates that the individual has high self-efficacy regarding their illness and believes they can achieve their goals."
Medication Adherence | 10 weeks
  The Medication Adherence Report Scale (MARS), developed by Horne and Hankins (2001), can be adapted based on disease type. The scale requires participants to indicate the frequency of occurrence for 5 specific statements in themselves. The scoring uses a Likert-type scale where: 5=never, 4=rarely, 3=sometimes, 2=often, and 1=always. The total test score is obtained by summing the scores from all items. The minimum possible score on the scale is 5, and the maximum is 25. Higher scores indicate compliance, while lower scores suggest non-compliance.
Sleep Quality | 10 weeks
  PSQI is developed by Buysse et al. in 1989, this scale is used to assess sleep quality and identify factors contributing to sleep disorders. Its validity and reliability for our country were established by Ağargün et al. The scale consists of 18 scored items grouped into 7 component scores, with each item rated on a 0-3 scale. The components are:
  Subjective Sleep Quality Sleep Latency Sleep Duration Habitual Sleep Efficiency Sleep Disturbances Use of Sleep Medication Daytime Dysfunction
  The total scale score is calculated by summing the seven component scores. A total score of 5 or higher indicates poor sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: AYLA DEMİRTAŞ, Associate Professor, Study Director — UNIVERSITY OF HEALTH SCIENCES GULHANE FACULTY OF NURSING
Locations (1):
- Gulhane Training and Research Hospital, Ankara, KEÇİÖREN, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No